CLINICAL TRIAL: NCT05451238
Title: Developing a Computerized Testing System for Measuring Motor and Sensory Integrative Functions in School-aged Children With Intellectual Disabilities
Brief Title: A Computerized Testing System for Measuring Motor and Sensory Integrative Functions in Children
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KMUHIRB-SV(II)-20190087
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Intellectual Disability
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Assessment of the motor and sensory integrative functions (MSI) is a key component of an overall health and functional evaluation for school-aged children with intellectual disabilities (ID). The ability of students with ID to perform age-appropriate motor tasks and adaptive behaviors (end product of sensory integration) can help determine the long-term effects of special education curriculum/interventions and the quality of an overall school-based rehabilitation program.We will develop item banks for 3 core domains of MSI (i.e., gross motor, fine motor, and sensory integration) for school-aged children with ID. About 200-250 participants will be recruited.

DETAILED DESCRIPTION:
Assessment of the motor and sensory integrative functions (MSI) is a key component of an overall health and functional evaluation for school-aged children with intellectual disabilities (ID). The ability of students with ID to perform age-appropriate motor tasks and adaptive behaviors (end product of sensory integration) can help determine the long-term effects of special education curriculum/interventions and the quality of an overall school-based rehabilitation program.

However, several challenges exist in measuring MSI for school-aged children with ID. First, most measures of MSI vary in content (domains), causing difficulty in the selection of relevant MSI measures. Second, most measures of MSI lack robust evidence of psychometric properties (e.g., reliability and responsiveness). Third, the minimal important difference (MID) and minimal detectable change (MDC) of most MSI measures for ID are largely unknown, which limits the interpretation of change scores in schools and clinical settings. Fourth, most MSI measures are time-consuming to administer, placing a burden of administration on both teachers/therapists and children. Finally, all the measures were developed in western countries and their use has not yet been validated for ID populations in Taiwan. An efficient and in-depth understanding of the students' motor and sensory integrative functions can help the school teachers implementing appropriate curriculum, monitoring the progress, managing the classroom, and further enhancing the overall learning for school-aged students with ID. A validated and convenient computerized testing system is urgently needed.

The Rasch model is useful in developing precise measures. Furthermore, a computerized adaptive testing (CAT) system can provide efficient measurements. Therefore, in this 3-year project, we will develop a Computerized Testing system for measuring Motor and Sensory Integrative Functioning in School-aged Children with Intellectual Disabilities (MSI-ID) to overcome the aforementioned challenges. We will determine whether the MSI-ID is efficient and psychometrically robust.

Method: We will develop item banks for 3 core domains of MSI (i.e., gross motor, fine motor, and sensory integration) for school-aged children with ID. We will select the 3 domains based on both core elements of a child's overall function and priorities of caregivers/teachers as determined in our preliminary study. We will construct 100 items for each domain based on focus group interviews of teachers / caregivers of students with ID and therapists, related theories and assessments, and suggestions from the experts. Then we will administer each item on 100 school-aged children with various levels of ID severity and age.

ELIGIBILITY:
Inclusion Criteria:

1. ages between 6 and 15 years; (2) a diagnosis of ID determined by the board-certified physicians at local designated hospitals according to the standards put forth by the International Classification of Diseases, 10th revision, clinical modification (ICD-10 codes); and (3) absence of serious emotional , behavioral disturbances or any other major disease affecting premorbid sensory processing and motor functions (e.g., muscular dystrophy).

Exclusion Criteria:

* None

Ages: 6 Years to 15 Years | Sex: All
Age Groups: Child
Study Population: school-aged children with different level of intellectual disabilities
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
BOT-2 | Baseline (pretest)
  The BOT-2 assesses proficiency in four motor-area composites: fine manual control composite, manual coordination composite, body coordination composite, and strength and agility composite. The average age-adjusted scale scores for subtests are 15 (S.D. = 5), whereas composites are derived by summing the subtest scale scores and converting them to a quotient with a mean of 100 and a S.D. of 15.
Jebsen-Taylor Hand Function Test | Baseline (pretest)
  The JTHFT is a quick and reliable measure of hand functioning incorporating 7 simulated tasks of activities of daily living (ADL).The tasks are: stacking, simulated page-turning, simulated feeding, picking up small objects, lifting large and lightweight object, lifting heavy object, and writing (copying). All tasks were timed and three scores were generated. A JTHFT- object score was the total time (seconds) taken to perform all 6 tasks except for writing for dominant and non-dominant hand, respectively. A JTHFT- writing score was the time spent (seconds) to complete a writing task for the dominant hand. Excellent reliabilities was reported in adults and typically developing children, and this assessment has also been utilized to exam the uni-manual capabilities in children with cerebral palsy and other motor dysfunctions
TVPS-4 | Baseline (pretest)
  The TVPS-4 is a motor-free and individually administered test to evaluate the comprehensive visual perceptual functions for individuals aged 5-21. The TVPS-4 comprised 7 tests: visual discrimination, visual memory, spatial relationship, form constancy, sequential memory, visual figure- ground, and visual closure. The TVPS-4 has excellent reliabilities evidence and concurrent validities with other similar tests
Sensory Profile | Baseline (pretest)
  The SP is a parent report measure of behaviors associated with abnormal responses to sensory stimuli for children 5-10 years of age. The SP consists of 125 items grouped into three main sections: Sensory Processing, Modulation, and Behavioral and Emotional Responses. Items are scored from always (1) to never (5), with higher scores indicating more impairment. The total score of each section is the best indicator of overall sensory dysfunction. The SP provides published cut-off scores. Scores at or above the mean are considered ''typical''; scores of 1 standard deviation below the mean for the typical reference sample are reported as a ''probable difference'', and scores at 2 standard deviations below the mean for the typical reference sample are reported as a ''definite difference''.
Vineland Adaptive Behavior Scale-Chinese Version | Baseline (pretest)
  The VABS-C was the Chinese version of the Vineland Adaptive Behavior Scale23 and was used in individuals aged 0 to 18 years-11 months. This assessment measures age-related adaptive skills essential for personal and social competencies. This 577-item measure included four domains: motor skills (gross, fine), communication (written, expressive, receptive,), daily living skills (community domestic, personal,), and socialization skills (coping skills, interpersonal relationships, play and leisure time)

CONTACTS AND LOCATIONS:
Overall Officials: Yee-Pay Wuang, PhD, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Dept of Occupational Therapy, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Haley SM, Ni P, Dumas HM, Fragala-Pinkham MA, Hambleton RK, Montpetit K, Bilodeau N, Gorton GE, Watson K, Tucker CA. Measuring global physical health in children with cerebral palsy: illustration of a multidimensional bi-factor model and computerized adaptive testing. Qual Life Res. 2009 Apr;18(3):359-70. doi: 10.1007/s11136-009-9447-5. Epub 2009 Feb 17. PMID 19221892
- See also: Measuring global physical health in children with cerebral palsy: illustration of a multidimensional bi-factor model and computerized adaptive testing. — https://pubmed.ncbi.nlm.nih.gov/19221892/